CLINICAL TRIAL: NCT06810934
Title: A Phase 1/2A, Randomized Study of a T Follicular Helper (TFH)-Targeting Genetic Vaccine Strategy Designed to Induce Broad, Durable Immune Responses
Acronym: CONTENDER
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kara Chew (Other)
Collaborators: University of California, San Francisco (Other); University of California, Davis (Other); Tendel Therapies, Inc. (Unknown); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Kara Chew, Associate Professor of Medicine, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 23-001884; 1U01AI172800-01A1 (NIH)
Record Dates: First submitted 2024-10-09; First posted 2025-02-06 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-07

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2; Vaccine; Adjuvant; Virus; RNA Virus Infections; Prevention; Immunogenicity; Immunity; Viral infection; Coronavirus Infection; Infection; Coronavirus Infections
MeSH Terms: conditions — COVID-19; Virus Diseases; RNA Virus Infections; Coronavirus Infections; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- Dose Cohort 1, Arm 1A (Experimental): Intervention: CoTend-s3BXBB (SARS2-17032) Dose: 1x10^6 vp (0.5mL) IM once
  Interventions: Biological: CoTend-s3BXBB (SARS2-17032)
- Dose Cohort 1, Arm 1B (Experimental): Intervention: CoTend-BXBB (SARS2-30404) Dose: 1x10^6 vp (0.5mL) IM once
  Interventions: Biological: CoTend-BXBB (SARS2-30404)
- Dose Cohort 2, Arm 2A (Experimental): Intervention: CoTend-s3BXBB (SARS2-17032) Dose: 1x10^7 vp (0.5mL) IM once
  Interventions: Biological: CoTend-s3BXBB (SARS2-17032)
- Dose Cohort 2, Arm 2B (Experimental): Intervention: CoTend-BXBB (SARS2-30404) Dose: 1x10^7 vp (0.5mL) IM once
  Interventions: Biological: CoTend-BXBB (SARS2-30404)
- Dose Cohort 3, Arm 3A (Experimental): Intervention: CoTend-s3BXBB (SARS2-17032) Dose: 1x10^8 vp (0.5mL) IM once
  Interventions: Biological: CoTend-s3BXBB (SARS2-17032)
- Dose Cohort 3, Arm 3B (Experimental): Intervention: CoTend-BXBB (SARS2-30404) Dose: 1x10^8 vp (0.5mL) IM once
  Interventions: Biological: CoTend-BXBB (SARS2-30404)
- Dose Cohort 4, Arm 4A (Experimental): Intervention: CoTend-s3BXBB (SARS2-17032) Dose: 1x10^9 vp (0.5mL) IM once
  Interventions: Biological: CoTend-s3BXBB (SARS2-17032)
- Dose Cohort 4, Arm 4B (Experimental): Intervention: CoTend-BXBB (SARS2-30404) Dose: 1x10^9 vp (0.5mL) IM once
  Interventions: Biological: CoTend-BXBB (SARS2-30404)
- Dose Cohort 5, Arm 5A (Experimental): Intervention: CoTend-s3BXBB (SARS2-17032) Dose: 1x10^10 vp (0.5mL) IM once
  Interventions: Biological: CoTend-s3BXBB (SARS2-17032)
- Dose Cohort 5, Arm 5B (Experimental): Intervention: CoTend-BXBB (SARS2-30404) Dose: 1x10^10 vp (0.5mL) IM once
  Interventions: Biological: CoTend-BXBB (SARS2-30404)
- Dose Cohort 6, Arm 6A (Experimental): Intervention: CoTend-s3BXBB (SARS2-17032) Dose: 1x10^9 vp (0.5mL) IM once
  Interventions: Biological: CoTend-s3BXBB (SARS2-17032)
- Dose Cohort 6, Arm 6B (Experimental): Intervention: CoTend-BXBB (SARS2-30404) Dose: 1x10^9 vp (0.5mL) IM once
  Interventions: Biological: CoTend-BXBB (SARS2-30404)
- Dose Cohort 6, Arm 6C (Placebo Comparator): Intervention: Placebo (normal saline) Dose: 0.5mL IM once
  Interventions: Biological: Placebo
- Dose Cohort 7, Arm 7A (Experimental): Intervention: CoTend-s3BXBB (SARS2-17032) Dose: 1x10^10 vp (0.5mL) IM once
  Interventions: Biological: CoTend-s3BXBB (SARS2-17032)
- Dose Cohort 7, Arm 7B (Experimental): Intervention: CoTend-BXBB (SARS2-30404) Dose: 1x10^10 vp (0.5mL) IM once
  Interventions: Biological: CoTend-BXBB (SARS2-30404)
- Dose Cohort 7, Arm 7C (Placebo Comparator): Intervention: Placebo (normal saline) Dose: 0.5mL IM once
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CoTend-BXBB (SARS2-30404) — Ad35-vectored SARS-CoV-2 RBD (XBB.1.5) vaccine
  Arms: Dose Cohort 1, Arm 1B; Dose Cohort 2, Arm 2B; Dose Cohort 3, Arm 3B; Dose Cohort 4, Arm 4B; Dose Cohort 5, Arm 5B; Dose Cohort 6, Arm 6B; Dose Cohort 7, Arm 7B
Biological: CoTend-s3BXBB (SARS2-17032) — Ad35-vectored s3-SARS-CoV-2 RBD (XBB.1.5) vaccine
  Arms: Dose Cohort 1, Arm 1A; Dose Cohort 2, Arm 2A; Dose Cohort 3, Arm 3A; Dose Cohort 4, Arm 4A; Dose Cohort 5, Arm 5A; Dose Cohort 6, Arm 6A; Dose Cohort 7, Arm 7A
Biological: Placebo — Sterile sodium chloride 0.9% for injection, preservative free
  Arms: Dose Cohort 6, Arm 6C; Dose Cohort 7, Arm 7C

SUMMARY:
The goal of this clinical trial is to test two investigational COVID-19 booster vaccines, called CoTend-s3BXBB and CoTend-BXBB, in healthy volunteers ages 40-64. The CoTend-s3BXBB vaccine includes a component called "s3", which was designed to improve the body's response to the vaccine. CoTend-BXBB is the same vaccine without s3.

The main questions the study aims to answer are: 1) Is the investigational vaccine safe? 2) Does "s3" lead to bigger, broader, and longer-lasting responses to the vaccine?

5 different doses of the vaccines will be studied. Participants will receive a single dose of either CoTend-s3BXBB, CoTend-BXBB, or placebo. Participants will be monitored for side effects. Saliva, nasal, and blood samples will be collected and immune responses to the vaccine will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals 40 - 64 years of age
2. Received at least two doses of a COVID-19 mRNA vaccine (Moderna or Pfizer) > 120 days before study entry
3. Nasal SARS-CoV-2 negative by molecular (polymerase chain reaction, PCR) testing at screening
4. The following laboratory criteria must be met at screening:

   1. Total white blood cell (WBC) count > 3500 cells/mm3
   2. Absolute neutrophil count (ANC) > 1500 cells/mm3
   3. Hemoglobin > 13.5 g/dL if male sex and > 12.0 g/dL if female sex
   4. Platelet count > 140,000/uL
   5. Estimated creatinine clearance (CrCl) > 50 mL/min by Cockroft-Gault equation
   6. Total bilirubin ≤ 1.1x upper limit of normal (ULN)
   7. Aspartate aminotransferase (AST) ≤ 1.3x ULN
   8. Alanine aminotransferase (ALT) ≤ 1.3x ULN
5. Individuals of reproductive potential must have a negative serum or urine beta-human chorionic gonadotropin (ß-HCG) test at screening and within 48 hours prior to entry.

   Reproductive potential is defined as:
   * Participants who have reached menarche
   * Participants who have not been post-menopausal for at least 12 consecutive months with follicle-stimulating hormone (FSH) ≥40 IU/mL or 24 consecutive months if an FSH is not available
   * Participants who have not undergone surgical contraception (e.g., hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or bilateral salpingectomy) NOTE: Participants who have undergone bilateral tubal ligation within the 24 weeks prior to screening are considered to be of reproductive potential and, if participating in sexual activity that could lead to pregnancy, contraception is required as per 5.2.2 exclusion criterion 2.
6. Able and willing to provide informed consent

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria are met:

1. Pregnant or breastfeeding
2. For participants capable of becoming pregnant and engaging in sexual activity that can lead to pregnancy, unwillingness to use contraception during participation in the study. For participants capable of becoming pregnant, two of the following forms of contraception are required through 30 days following administration of study intervention, one of which must be a barrier method:

   1. Condoms (male or female) with or without a spermicidal agent
   2. Diaphragm or cervical cap with spermicide
   3. Intrauterine device (IUD)
   4. Hormone-based contraceptive such as oral birth control pills
3. Known close contact with anyone with confirmed SARS-CoV-2 infection (defined as positive SARS-CoV-2 nucleic acid or antigen testing by laboratory-based or home self-test) within 2 weeks prior to expected study entry
4. Plan to receive a non-study SARS-CoV-2 vaccine within 8 weeks after study entry
5. HIV infection
6. Hepatitis B core antibody or hepatitis B surface antigen positive at screening
7. Current active hepatitis C. Participants must be hepatitis C virus (HCV) antibody negative or have evidence of cleared HCV infection. If the participant is HCV antibody positive or indeterminate, an unquantifiable HCV RNA result (below lower limit of quantification, either target detected or target not detected) within 42 days prior to study entry is required. Those who are currently receiving HCV antiviral therapy or those who have received HCV treatment in the last 3 months prior to study entry will be excluded.
8. History of cirrhotic liver disease
9. History of thrombosis with thrombocytopenia syndrome (TTS), immune thrombocytopenia, thromboembolic events, capillary leak syndrome, other thrombotic disease or known increased risk of thrombosis due to genetic disorders or malignancy
10. History of or active autoimmune disease that has required systemic immunosuppressive or immunomodulatory therapy
11. History of myocarditis, pericarditis, or myopericarditis
12. Potential myocarditis or pericarditis identified at screening, defined as high-sensitivity troponin I (hsTnI) > ULN or 12-lead ECG compatible with pericarditis WITH compatible symptoms (regardless of troponin I level) at screening
13. History of Guillain-Barré syndrome
14. History of coagulopathy or bleeding disorder considered a contraindication to intramuscular injection or phlebotomy
15. Symptomatic acute or chronic illness requiring ongoing medical or surgical care, including requirement for new medications, in the past 3 months. Transient illnesses or injuries that are resolved prior to screening are not exclusionary. Minor adjustments in stable therapy for chronic conditions such as hypertension are not exclusionary. Use of over-the-counter medications for any acute or chronic illness is also not exclusionary.
16. Serious medical or psychiatric illness that, in the opinion of the site investigator, would interfere with the ability to adhere to study requirements or to give informed consent
17. Treatment with systemic immunosuppressive or immunomodulatory drugs, and/or exposure to any immunosuppressive/immunomodulatory drug in the 30 days prior to study entry (e.g. corticosteroid therapy equal to or exceeding a dose of 20 mg/day of prednisone for more than 10 days, interleukins, interferons, methotrexate, rituximab, and cancer chemotherapy). Use of topical, inhaled, intra-articular, or nasal steroid use is not exclusionary.
18. Active malignancy or history of malignancy within the 4 years prior to study entry. Non-melanoma skin cancers (such as basal or squamous cell skin cancers) and non-invasive cervical or anal intraepithelial lesions are not exclusionary.
19. History of solid organ or hematopoietic stem cell transplantation
20. History of primary immunodeficiency disorder
21. Ongoing complications or morbidity associated with prior diagnoses of malignancies requiring continued medical or surgical intervention. Chronic stable complications or morbidity not requiring new medications or other medical or surgical intervention in the past 3 months are not exclusionary.
22. Administration or planned administration of blood products or licensed non-SARS-CoV-2 vaccines <14 days prior to or within 14 days after study entry
23. Receipt of any antibody-based therapy (investigational or approved) for prophylaxis or treatment of COVID-19 in the preceding 6 months
24. Receipt of immunoglobulin therapy in the year prior to study entry or scheduled or anticipated immunoglobulin administration during the study period.
25. Prior receipt of any non-mRNA SARS-CoV-2 vaccine
26. Receipt of any SARS-CoV-2 vaccination in the 120 days prior to study entry
27. Documented SARS-CoV-2 infection in the 120 days prior to study entry
28. History of anaphylaxis, urticaria, or other significant adverse reaction requiring medical intervention (medications requiring a prescription or surgical intervention) after receipt of a vaccine or intervention that includes one or more of the same components contained in the study product
29. Have participated in an interventional clinical study within 28 days prior to screening (based on medical history interview) or plans to do so while participating in this study
30. Any clinical concerns as determined by the investigator that might affect the potential participant's safety in the study.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of solicited local reactogenicity adverse events (AEs) within 7 days after dosing. | 7 days
  Number of participants with solicited local reactogenicity AEs (injection site pain, erythema, or swelling) within 7 days after dosing. An AE is any untoward medical occurrence in a clinical investigation of a patient administered a pharmaceutical product and that does not necessarily have a causal relationship with the treatment.
Frequency of solicited systemic reactogenicity AEs within 7 days after dosing. | 7 days
  Number of participants with solicited systemic reactogenicity AEs (malaise, participant-measured body temperature, fatigue, headache, chills, nausea, muscle aches/pain, joint pain) within 7 days after dosing.
Frequency of unsolicited AEs within 28 days after dosing. | 28 days
  Number of participants with unsolicited AEs within 28 days after dosing. Unsolicited AEs are AEs that were not pre-defined as solicited.
Frequency of serious adverse events (SAEs) within 28 days after dosing. | 28 days
  Number of participants with an SAE within 28 days after dosing. An SAE is defined as any adverse event that results in any of the following outcomes: death during a period of surveillance defined by the protocol, a life-threatening adverse experience, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect. The following are also considered SAEs for this study: severe COVID-19, defined as COVID-19 requiring hospitalization or supplemental oxygen, myocarditis or pericarditis within 6 weeks of study vaccination, and acute or new onset thrombosis or thromboembolism within 60 days of vaccination.
Frequency of adverse events of special interest (AESIs) within 28 days after dosing. | 28 days
  Number of participants with AESIs. AESIs defined as: thrombotic or thromboembolic events, thrombosis with thrombocytopenia syndrome, immune thrombocytopenia, or capillary leak syndrome occurring within 60 days; new thrombocytopenia <150 x 10^9/L or below the lower laboratory limit of normal or worsening in grade of thrombocytopenia within 60 days after study vaccination; new D-dimer elevation >2000 ng/mL within 60 days; laryngospasm, bronchospasm, or anaphylaxis assessed as at least possibly related; generalized urticaria assessed as related; any other grade allergic/ hypersensitivity reaction within 7 days; any ulceration, abscess, or necrosis at injection site assessed as possibly related; myocarditis or pericarditis occurring within 6 weeks; new diagnosis of Guillain-Barré syndrome occurring within 60 days; any new or worsened immune mediated medical condition; grade 3+ lab abnormality for which there is a reasonable possibility of causal relationship to study treatment.
Frequency of medically attended adverse events (MAAEs) within 28 days after dosing. | 28 days
  Number of participants with MAAEs (MAAE defined as an AE resulting in a hospitalization, emergency room visit, or otherwise unscheduled visit with medical personnel for any reason) within 28 days after dosing.
Geometric mean titers (GMTs) of serum anti-XBB.1.5 neutralizing antibodies (NAb) through week 8. | 8 weeks
  Serum anti-XBB.1.5 NAb GMT
Proportion of participants achieving serum anti-XBB.1.5 NAb titers of 1:250 or better through week 8. | 8 weeks
  Proportion of participants achieving serum anti-XBB.1.5 NAb titers of 1:250 or better
Geometric mean fold rise (GMFR) from pre-dose to week 8 in serum anti-XBB.1.5 NAb responses. | Pre-dose to 8 weeks
  Geometric mean fold rise (GMFR) in serum anti-XBB.1.5 NAb levels

SECONDARY OUTCOMES:
Serum anti-D614G NAb GMTs through week 8. | 8 weeks
  Serum anti-D614G NAb GMTs
Serum anti-JN.1* NAb GMTs through week 8. | 8 weeks
  Serum anti-JN.1* NAb GMTs (*the most relevant SARS-CoV-2 variant at the time of analysis will be evaluated)
Proportion of participants achieving anti-D614G NAb titers of 1:250 or better through week 8. | 8 weeks
  Proportion of participants achieving anti-D614G NAb titers of 1:250 or better
Proportion of participants achieving anti-JN.1* NAb titers of 1:250 or better through week 8. | 8 weeks
  Proportion of participants achieving serum anti-JN.1* NAb GMTs of 1:250 or better (*the most relevant SARS-CoV-2 variant at the time of analysis will be evaluated).
GMFR from pre-dose to week 8 in serum anti-D614G NAb responses. | Pre-dose to 8 weeks
  GMFR in serum anti-D614G NAb responses
GMFR from pre-dose to week 8 in serum anti-JN.1* NAb responses. | Pre-dose to 8 weeks
  GMFR in serum anti-JN.1* NAb responses (*the most relevant SARS-CoV-2 variant at the time of analysis will be evaluated).
Serum anti-XBB.1.5 RBD IgG binding antibody (bAb) GMTs through week 8. | 8 weeks
  Serum anti-XBB.1.5 RBD IgG bAb GMTs
Serum anti-XBB.1.5 RBD IgA binding antibody GMTs through week 8. | 8 weeks
  Serum anti-XBB.1.5 RBD IgA bAb GMTs
Serum anti-D614G RBD IgG binding antibody (bAb) GMTs through week 8. | 8 weeks
  Serum anti-D614G RBD IgG bAb GMTs.
Serum anti-D614G RBD IgA binding antibody (bAb) GMTs through week 8. | 8 weeks
  Serum anti-D614G RBD IgA bAb GMTs through week 8.
Serum anti-JN.1* RBD IgG binding antibody (bAb) GMTs through week 8. | 8 weeks
  Serum anti-JN.1* RBD IgG bAb GMTs (*the most relevant SARS-CoV-2 variant at the time of analysis will be evaluated)
Serum anti-JN.1* RBD IgA binding antibody (bAb) GMTs through week 8. | 8 weeks
  Serum anti-JN.1* RBD IgA bAb GMTs (*the most relevant SARS-CoV-2 variant at the time of analysis will be evaluated)
Geometric mean fold rise (GMFR) from pre-dose to week 8 in serum anti-XBB.1.5 RBD IgG binding antibody responses. | Pre-dose to 8 weeks
Geometric mean fold rise (GMFR) from pre-dose to week 8 in serum anti-XBB.1.5 RBD IgA binding antibody responses. | Pre-dose to 8 weeks
Geometric mean fold rise (GMFR) from pre-dose to week 8 in serum anti-D614G RBD IgG binding antibody responses. | Pre-dose to 8 weeks
Geometric mean fold rise (GMFR) from pre-dose to week 8 in serum anti-D614G RBD IgA binding antibody responses. | Pre-dose to 8 weeks
Geometric mean fold rise (GMFR) from pre-dose to week 8 in serum anti-JN.1* RBD IgG binding antibody responses. | Pre-dose to 8 weeks
Geometric mean fold rise (GMFR) from pre-dose to week 8 in serum anti-JN.1* RBD IgA binding antibody responses. | Pre-dose to 8 weeks
Frequency of grade 3 or higher AEs through week 26 visit. | 26 weeks
  Number of participants with grade 3 or higher AEs through week 26 visit. Grade 3 AE is defined as severe symptoms causing inability to perform usual social and functional activities with intervention or hospitalization indicated. Grade 4 AE is defined as potentially life-threatening symptoms causing inability to perform basic self-care functions with intervention indicated to prevent permanent impairment, persistent disability, or death. All deaths related to an AE are classified as grade 5.
Frequency of SAEs through week 26 visit. | 26 weeks
  Number of participants with SAEs through week 26 visit.
Frequency of AESIs through week 26 visit. | 26 weeks
  Number of participants with AESIs through week 26 visit.
Frequency of MAAEs through week 26 visit. | 26 weeks
  Number of participants with MAAEs through week 26 visit
Frequency of SAEs through end of study visit | Through end of study visit (52 or 104 weeks)
  Number of participants with SAEs through their end of study visit
Frequency of AESIs through end of study visit | Through end of study visit (52 or 104 weeks)
  Number of participants with AESIs through their end of study visit
Frequency of MAAEs through end of study visit | Through end of study visit (52 or 104 weeks)
  Number of participants with MAAEs through their end of study visit
Fraction of RBD-specific CD4+ T cells through week 8. | 8 weeks
  Fraction of RBD-specific CD4+ T cells
Fraction of RBD-specific CD8+ T cells through week 8. | 8 weeks
  Fraction of RBD-specific CD8+ T cells
NAb GMTs through week 26. | 26 weeks
  Serum NAb GMTs
NAb GMTs through week 52. | 52 weeks
  Serum NAb GMTs
NAb GMTs through week 104. | 104 weeks
  Serum NAb GMTs
Binding Ab GMTs through week 26. | 26 weeks
  Serum binding Ab GMTs
Binding Ab GMTs through week 52. | 52 weeks
  Serum binding Ab GMTs
Binding Ab GMTs through week 104. | 104 weeks
  Serum binding Ab GMTs
Proportion of participants achieving NAb titers of 1:250 or better through week 26. | 26 weeks
  Proportion of participants achieving serum NAb titers of 1:250 or better
Proportion of participants achieving NAb titers of 1:250 or better through week 52. | 52 weeks
  Proportion of participants achieving serum NAb titers of 1:250 or better
Proportion of participants achieving NAb titers of 1:250 or better through week 104. | 104 weeks
  Proportion of participants achieving serum NAb titers of 1:250 or better
GMFR of NAb titers from pre-dose through week 26. | Pre-dose to 26 weeks
  GMFR of serum NAb titers
GMFR of NAb titers from pre-dose through week 52. | Pre-dose to 52 weeks
  GMFR of serum NAb titers
GMFR of NAb titers from pre-dose through week 104. | Pre-dose to 104 weeks
  GMFR of serum NAb titers
GMFR of binding Ab titers from pre-dose through week 26. | Pre-dose to 26 weeks
GMFR of binding Ab titers from pre-dose through week 52. | Pre-dose to 52 weeks
GMFR of binding Ab titers from pre-dose through week 104. | Pre-dose to 104 weeks
Fraction of RBD-specific CD4+ T cells through week 26. | 26 weeks
  Fraction of RBD-specific CD4+ T cells
Fraction of RBD-specific CD4+ T cells through week 52. | 52 weeks
  Fraction of RBD-specific CD4+ T cells
Fraction of RBD-specific CD4+ T cells through week 104. | 104 weeks
  Fraction of RBD-specific CD4+ T cells
Fraction of RBD-specific CD8+ T cells through week 26. | 26 weeks
  Fraction of RBD-specific CD8+ T cells
Fraction of RBD-specific CD8+ T cells through week 52. | 52 weeks
  Fraction of RBD-specific CD8+ T cells
Fraction of RBD-specific CD8+ T cells through week 104. | 104 weeks
  Fraction of RBD-specific CD8+ T cells

CONTACTS AND LOCATIONS:
Overall Officials: Kara Chew, MD, MS, Principal Investigator — University of California, Los Angeles; Steven Deeks, MD, Principal Investigator — University of California, San Francisco; Dennis Hartigan-O'Connor, MD, PhD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - UCLA Westwood, Los Angeles, California
  - UCSF Community and Clinical Research Center, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
De-identified data.
Time Frame: After completion of the study analyses and publications.
Access Criteria: There will be a managed access process with requirement of a data use agreement.

REFERENCES:
- [Background] Bowen JE, Park YJ, Stewart C, Brown JT, Sharkey WK, Walls AC, Joshi A, Sprouse KR, McCallum M, Tortorici MA, Franko NM, Logue JK, Mazzitelli IG, Nguyen AW, Silva RP, Huang Y, Low JS, Jerak J, Tiles SW, Ahmed K, Shariq A, Dan JM, Zhang Z, Weiskopf D, Sette A, Snell G, Posavad CM, Iqbal NT, Geffner J, Bandera A, Gori A, Sallusto F, Maynard JA, Crotty S, Van Voorhis WC, Simmerling C, Grifantini R, Chu HY, Corti D, Veesler D. SARS-CoV-2 spike conformation determines plasma neutralizing activity elicited by a wide panel of human vaccines. Sci Immunol. 2022 Dec 23;7(78):eadf1421. doi: 10.1126/sciimmunol.adf1421. Epub 2022 Dec 23. PMID 36356052
- [Background] De Boer RJ, Perelson AS. How Germinal Centers Evolve Broadly Neutralizing Antibodies: the Breadth of the Follicular Helper T Cell Response. J Virol. 2017 Oct 27;91(22):e00983-17. doi: 10.1128/JVI.00983-17. Print 2017 Nov 15. PMID 28878083
- [Background] Wang Q, Iketani S, Li Z, Liu L, Guo Y, Huang Y, Bowen AD, Liu M, Wang M, Yu J, Valdez R, Lauring AS, Sheng Z, Wang HH, Gordon A, Liu L, Ho DD. Alarming antibody evasion properties of rising SARS-CoV-2 BQ and XBB subvariants. Cell. 2023 Jan 19;186(2):279-286.e8. doi: 10.1016/j.cell.2022.12.018. Epub 2022 Dec 14. PMID 36580913
- [Background] Havervall S, Marking U, Svensson J, Greilert-Norin N, Bacchus P, Nilsson P, Hober S, Gordon M, Blom K, Klingstrom J, Aberg M, Smed-Sorensen A, Thalin C. Anti-Spike Mucosal IgA Protection against SARS-CoV-2 Omicron Infection. N Engl J Med. 2022 Oct 6;387(14):1333-1336. doi: 10.1056/NEJMc2209651. Epub 2022 Sep 14. No abstract available. PMID 36103621
- [Background] Balachandran H, Phetsouphanh C, Agapiou D, Adhikari A, Rodrigo C, Hammoud M, Shrestha LB, Keoshkerian E, Gupta M, Turville S, Christ D, King C, Sasson SC, Bartlett A, Grubor-Bauk B, Rawlinson W, Aggarwal A, Stella AO, Klemm V, Mina MM, Post JJ, Hudson B, Gilroy N, Konecny P, Ahlenstiel G, Dwyer DE, Sorrell TC, Kelleher A, Tedla N, Lloyd AR, Martinello M, Bull RA; COSIN Study Group. Maintenance of broad neutralizing antibodies and memory B cells 1 year post-infection is predicted by SARS-CoV-2-specific CD4+ T cell responses. Cell Rep. 2022 Feb 8;38(6):110345. doi: 10.1016/j.celrep.2022.110345. Epub 2022 Jan 19. PMID 35090598
- [Background] Fuchs JD, Bart PA, Frahm N, Morgan C, Gilbert PB, Kochar N, DeRosa SC, Tomaras GD, Wagner TM, Baden LR, Koblin BA, Rouphael NG, Kalams SA, Keefer MC, Goepfert PA, Sobieszczyk ME, Mayer KH, Swann E, Liao HX, Haynes BF, Graham BS, McElrath MJ; NIAID HIV Vaccine Trials Network. Safety and Immunogenicity of a Recombinant Adenovirus Serotype 35-Vectored HIV-1 Vaccine in Adenovirus Serotype 5 Seronegative and Seropositive Individuals. J AIDS Clin Res. 2015 May;6(5):461. doi: 10.4172/2155-6113.1000461. Epub 2015 May 23. PMID 26587311
- [Background] Nwanegbo E, Vardas E, Gao W, Whittle H, Sun H, Rowe D, Robbins PD, Gambotto A. Prevalence of neutralizing antibodies to adenoviral serotypes 5 and 35 in the adult populations of The Gambia, South Africa, and the United States. Clin Diagn Lab Immunol. 2004 Mar;11(2):351-7. doi: 10.1128/cdli.11.2.351-357.2004. PMID 15013987
- [Background] Qu P, Faraone JN, Evans JP, Zheng YM, Yu L, Ma Q, Carlin C, Lozanski G, Saif LJ, Oltz EM, Gumina RJ, Liu SL. Durability of Booster mRNA Vaccine against SARS-CoV-2 BA.2.12.1, BA.4, and BA.5 Subvariants. N Engl J Med. 2022 Oct 6;387(14):1329-1331. doi: 10.1056/NEJMc2210546. Epub 2022 Sep 7. No abstract available. PMID 36069925
- [Background] Gilboa M, Regev-Yochay G, Mandelboim M, Indenbaum V, Asraf K, Fluss R, Amit S, Mendelson E, Doolman R, Afek A, Freedman LS, Kreiss Y, Lustig Y. Durability of Immune Response After COVID-19 Booster Vaccination and Association With COVID-19 Omicron Infection. JAMA Netw Open. 2022 Sep 1;5(9):e2231778. doi: 10.1001/jamanetworkopen.2022.31778. PMID 36107426
- [Background] Chen Y, Tong P, Whiteman NB, et al. Differential antibody dynamics to SARS-CoV-2 infection and vaccination. bioRxiv 2021:2021.09.09.459504.
- [Background] Planas D, Veyer D, Baidaliuk A, Staropoli I, Guivel-Benhassine F, Rajah MM, Planchais C, Porrot F, Robillard N, Puech J, Prot M, Gallais F, Gantner P, Velay A, Le Guen J, Kassis-Chikhani N, Edriss D, Belec L, Seve A, Courtellemont L, Pere H, Hocqueloux L, Fafi-Kremer S, Prazuck T, Mouquet H, Bruel T, Simon-Loriere E, Rey FA, Schwartz O. Reduced sensitivity of SARS-CoV-2 variant Delta to antibody neutralization. Nature. 2021 Aug;596(7871):276-280. doi: 10.1038/s41586-021-03777-9. Epub 2021 Jul 8. PMID 34237773